CLINICAL TRIAL: NCT05418049
Title: Evaluating the Neurophysiologic and Clinical Effects of Single-Dose Baclofen, Roflumilast, Memantine, and Placebo in Fragile X Syndrome
Brief Title: Evaluating the Neurophysiologic and Clinical Effects of Single Dose Drug Challenge
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-0202; U54HD104461 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Baclofen; Memantine; Roflumilast

STUDY DESIGN:
Intervention Model Description: This study was designed as a 4-intervention crossover, with all study participants receiving all possible interventions. These are placebo, baclofen, roflumilast, and memantine.
Masking Description: Quadruple masking (participant, care provider, investigator and outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Study Participants (Experimental): Participants received, in random order, a single dose of placebo, baclofen, roflumilast or memantine with a two-week washout period between doses.
  Interventions: Drug: Baclofen; Drug: Memantine; Drug: Roflumilast
- Control Study Participants (Placebo Comparator): Participants received, in random order, a single dose of placebo, baclofen, roflumilast or memantine with a two-week washout period between doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — 30mg - Supplied as 10mg and 20mg tablets
  Arms: Experimental Study Participants
Drug: Memantine — two 10 mg tablets
  Other Names: NAMENDA
  Arms: Experimental Study Participants
Drug: Roflumilast — 250 mcg capsule
  Other Names: DAILIRESP
  Arms: Experimental Study Participants
Drug: Placebo — Placebo pill
  Arms: Control Study Participants

SUMMARY:
The aim of this study is to utilize neurophysiologic assessments, behavioral measures and clinical measures to assess how much deficits associated with Fragile X Syndrome from pre-dose to post-dose using pharmacology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages 18-45, with FXS who completed the study entitled "Mechanisms and brain circuits underlying fragile X syndrome" (IRB # 2015-8425) or appropriate baseline measures through Biorepository (2013-7327).
* FXS is defined as full FMR1 mutations (>200 CGG repeats) confirmed by genetic testing.
* General good health as determined by physical exam, medical history and laboratory work up.
* Stanford Binet IQ <85
* Stable dosing of psychotropic drugs for at least 4 weeks.

Exclusion Criteria:

* Subjects with a history of intolerance to baclofen, roflumilast, or memantine will be excluded.
* Subjects will also be excluded if they have taken any investigational drug within 3 months, have a history of substance abuse or dependence within 6 months, or significant psychiatric or CNS neurological disease unrelated to FXS.
* Uncontrolled seizures or history of epilepsy with a seizure in the past 6 months
* Auditory or visual impairments that cannot be corrected based on visual and auditory screener benchmarks.
* Moderate to severe renal or hepatic impairment and determined by a study physician incorporating data from exam, medical history and laboratory value evaluation among other data points.
* Use of barbiturates, benzodiazepines, antiepileptics, or other GABAergic or glutamatergic modulators
* Current use of: Amifampridine, Butalbital, Codeine, Doxylamine, Ethanol, Hydrocodone, Isocarboxazid, Kava, Metoclopramide, Midazolam, Oxybate, Phenelzine, Promethazine, Thalidomide, Tranylcypromine, Trimethobenzamide, Erythromycin, Ketoconazole, Fluvoxamine, Enoxacin, and Cimetidine.
* Those taking other psychiatric medications must be on stable doses for 4 weeks before the baseline visit.
* Pregnancy or breast-feeding. For female subjects of child bearing potential, a urine pregnancy test will be performed.
* Potential subjects with a creatinine clearance < 50 mL/min will be excluded.
* Identified medical issues, inability to tolerate study procedures or study drug per the discretion of the Principal Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Change in EEG Relative Gamma Power | Pre-dose, 3-hour post-dose
  EEG relative gamma power at rest was calculated as the percent of power in the gamma frequencies relative to the sum of power in all frequency bands, averaged across electrodes, and calculated separately at pre-dose and post-dose timepoints. To assess the impact of drug, the pre-dose relative gamma power was subtracted from post-dose relative gamma power. Higher numbers indicate more relative gamma power post-dose; lower numbers indicate more relative gamma power pre-dose.

SECONDARY OUTCOMES:
Clinical Global Impressions-Improvement | Pre-dose, 3-hour post-dose
  The Clinical Global Impressions - Improvement (CGI-I) requires the clinician to assess how much the patient's illness has changed relative to pre-dose, from 1 (very much improved) to 7 (very much worse).
Clinical Global Impressions-Improvement-Caregiver | Pre-dose, 3-hour post-dose
  The CGI-I requires the caregiver to assess how much the patient's illness has changed relative to pre-dose, from 1 (very much improved) to 7 (very much worse).
Visual Analog Scale - Caregiver | Pre-dose, 3-hour post-dose
  The parent or caregiver will be asked to assess how much anxiety the participant is expressing on a line between two endpoints (no anxiety to worsened anxiety).

OTHER OUTCOMES:
Probabilistic Reversal Learning (PRL) | Pre-dose, 3-hour post-dose
  An examinee will be prompted to complete four different reversal learning tasks on a computer, each which had two phases: Acquisition and Reversal. Participants will be instructed to choose one of two identical stimuli positioned in different locations on the screen. Participant behavior will be reinforced on 80% of correct responses and on 20% of incorrect responses. During the acquisition phase, participants chose one of two stimulus locations until they identified the correct location on 8 of 10 consecutive trials. Then, they proceeded to the reversal phase in which the correct location is switched without warning, and participants had to identify the new correct location on 8 of 10 consecutive trials. Testing was discontinued if they did not reach criterion within 50 trials on either phase. Participants completed two practice tests to establish test comprehension. We computed total number of trials to reach criterion and number of errors after reversal.
NIH Cognitive Toolbox | 3-hour post-dose
  Computerized tasks comprised of 3 subtests where an examinee is shown a series of target stimuli, oral reading components, directional decision-making and picture vocabulary.
Expressive Language Sampling (ELS) | 3 hour post-dose
  An examinee will provide a sample of their spoken language while they create a narrative of a story. Participants were asked to tell the story of a wordless picture book "Frog Goes to Dinner." First the examiner showed the participant each page of the book at a 10 s interval per page. The examiner then asked the participant to tell the story page by page. The examiner utilized scripted prompts to encourage the participants to narrate the book with his/her own words. Digital audio-recorded samples were then de-identified and transferred to the at the UC Davis MIND Institute for transcription and analysis. The samples were transcribed using Systematic Analysis of Language Transcripts, 2018 Research Version software (SALT). The SALT program performs predetermined and customized analysis of text language files.
Test of Attentional Performance for Children (KiTAP) Test of Alertness | Pre-dose, 3-hour post-dose
  Computerized task where an examinee is required to push a key when a target stimulus is presented on the screen. Scores are presented as change in median reaction time (RT), in milliseconds.
Eye-tracking | Pre-dose, 3-hour post-dose
  An examinee will observe a series of pictures and videos on a computer screen where a video will capture gaze preference.

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Erickson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States